CLINICAL TRIAL: NCT06613503
Title: Testing the Effectiveness of the AI-Supporter in Reducing Urinary Tract Infections, Incontinence-associated Dermatitis and Caregiving Costs for Incontinence Patients
Brief Title: Effectiveness of the AI-Supporter in Reducing Urinary Tract Infections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CMUH113-REC3-109
Record Dates: First submitted 2024-09-18; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Incontinence; Urinary Tract Infection; Incontinence-associated Dermatitis; Cost-effectiveness
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Model Description: In this clinical trial, a parallel design is employed, where participants are randomly assigned to one of two groups: an experimental group and a control group. The experimental group will use the AI-supporter for excretion detection, cleaning, and drying processes, while the control group will use traditional diapers for care. The two groups will not cross over during the trial, meaning participants will remain in their assigned group throughout the study. This design allows for a direct comparison of the intervention's efficacy, with each group receiving a distinct form of care. The primary objective is to assess the effectiveness of the AI-supporter in reducing urinary tract infections and incontinence-associated dermatitis
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-supporter (Experimental): Participants will use the AI-supporter for excretion detection, cleaning, and drying processes.
  Interventions: Device: AI-supporter
- Traditional Diapers (No Intervention): Participants will use theTraditional Diapers for excretion detection, cleaning, and drying processes

INTERVENTIONS:
Device: AI-supporter — rticipants in the experimental group will use the AI-supporter, an intelligent excretion management robot. This device utilizes AI-driven visual recognition technology to automatically detect urine and feces, followed by a cleaning and drying process. When the AI-supporter detects excretion, it activates an automated sequence that washes, dries, and sanitizes the perineal area without requiring the caregiver to remove the diaper. The AI-supporter also records relevant data, such as the time, frequency, and weight of excretion, for further analysis. This intervention is designed to reduce the incidence of urinary tract infections (UTIs) and incontinence-associated dermatitis (IAD), as well as lessen the workload for caregivers
  Other Names: tradiational diapear
  Arms: AI-supporter

SUMMARY:
The "AI Supporter," an intelligent excretion management robot, leverages artificial intelligence-based vision recognition to autonomously detect and cleanse affected areas, followed by drying and changing the diaper, thereby reducing caregiver strain and enhancing care quality. This study aims to assess the efficacy of the "AI Supporter" in decreasing the incidence of urinary tract infections and incontinence-associated dermatitis among incontinent patients, in addition to exploring its cost-effectiveness.

Adopting an experimental (two groups) and longitudinal design, this research utilizes both convenience and random sampling strategies. The study anticipates recruiting 60 female subjects who have been confined to bed for more than three months with urinary and/or fecal incontinence. Participants will intermittently use the AI Supporter over a 14-day period. Measurement tools include routine urine analysis.

DETAILED DESCRIPTION:
Background: As Taiwan progresses medically, the aging demographic has become a significant challenge, leading to an escalation in the disabled population. The lack of caregiving manpower represents a critical bottleneck in the provision of long-term care. Diaper changing, a daily and labor-intensive task for caregivers, involves bending motions that pose a risk of musculoskeletal injuries. Consequently, the imperative development of automated caregiving technologies has emerged. The "AI Supporter," an intelligent excretion management robot, leverages artificial intelligence-based vision recognition to autonomously detect and cleanse affected areas, followed by drying and changing the diaper, thereby reducing caregiver strain and enhancing care quality.

Objective: This study aims to assess the efficacy of the "AI Supporter" in decreasing the incidence of urinary tract infections and incontinence-associated dermatitis among incontinent patients, in addition to exploring its cost-effectiveness.

Methods: Adopting an experimental (two groups) and longitudinal design, this research utilizes both convenience and random sampling strategies. Scheduled from November 2024 to October 2025 at a residential long-term care facility in Central Taiwan, the study anticipates recruiting 60 female subjects who have been confined to bed for more than three months with urinary and/or fecal incontinence. Participants will intermittently use the AI Supporter over a 14-day period. Measurement tools include routine urine analysis, incontinence-associated dermatitis rating scales, pressure sore assessments, skin pH measurements, caregiver hours, and cost analyses pertaining to diapers and the AI Supporter. The principal analytical method employed will be Generalized Estimating Equations (GEE), with statistical significance defined at p < 0.05.

Expected Outcomes: The AI Supporter is expected to significantly reduce the occurrence of urinary tract infections and incontinance-associated dermatitis in patients, concurrently alleviating caregiver workload and diminishing associated costs.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been bedridden for at least 3 months and have urinary and/or fecal incontinence.
* Female participants aged over 20 years old.
* Participants must be capable of wearing the AI-supporter device during the study period.

Exclusion Criteria:

* Participants with severe skin conditions unrelated to incontinence.
* Participants with current urinary tract infections or incontinence-associated dermatitis at the time of enrollment.
* Participants who are unable to provide informed consent or have a legal representative to do so.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
white blood cells | 14 days after intervention
  urine analysis
Bacterial count | 14 days after intervention
  urine analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kwo-Chen Lee, ph.D, Study Director — 011+886+4+22053366#7102
Locations (1):
- Rom A Master List, Extracted From This Organization'S Records., Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borchert K, Bliss DZ, Savik K, Radosevich DM. The incontinence-associated dermatitis and its severity instrument: development and validation. J Wound Ostomy Continence Nurs. 2010 Sep-Oct;37(5):527-35. doi: 10.1097/WON.0b013e3181edac3e. PMID 20736860
- [Background] Buckingham KW, Berg RW. Etiologic factors in diaper dermatitis: the role of feces. Pediatr Dermatol. 1986 Feb;3(2):107-12. doi: 10.1111/j.1525-1470.1986.tb00499.x. PMID 3513143
- [Background] Fader M, Clarke-O'Neill S, Cook D, Dean G, Brooks R, Cottenden A, Malone-Lee J. Management of night-time urinary incontinence in residential settings for older people: an investigation into the effects of different pad changing regimes on skin health. J Clin Nurs. 2003 May;12(3):374-86. doi: 10.1046/j.1365-2702.2003.00731.x. PMID 12709112
- [Background] Ferreira M, Abbade L, Bocchi SCM, Miot HA, Boas PV, Guimaraes HQCP. Incontinence-associated dermatitis in elderly patients: prevalence and risk factors. Rev Bras Enferm. 2020;73 Suppl 3:e20180475. doi: 10.1590/0034-7167-2018-0475. Epub 2020 Jul 13. English, Portuguese. PMID 32696899
- [Background] Francis K, Pang SM, Cohen B, Salter H, Homel P. Disposable Versus Reusable Absorbent Underpads for Prevention of Hospital-Acquired Incontinence-Associated Dermatitis and Pressure Injuries. J Wound Ostomy Continence Nurs. 2017 Jul/Aug;44(4):374-379. doi: 10.1097/WON.0000000000000337. PMID 28549048
- [Background] Gray M. Optimal management of incontinence-associated dermatitis in the elderly. Am J Clin Dermatol. 2010;11(3):201-10. doi: 10.2165/11311010-000000000-00000. PMID 20131923
- [Background] Hachem JP, Crumrine D, Fluhr J, Brown BE, Feingold KR, Elias PM. pH directly regulates epidermal permeability barrier homeostasis, and stratum corneum integrity/cohesion. J Invest Dermatol. 2003 Aug;121(2):345-53. doi: 10.1046/j.1523-1747.2003.12365.x. PMID 12880427
- [Background] Hahnel E, Blume-Peytavi U, Trojahn C, Kottner J. Associations between skin barrier characteristics, skin conditions and health of aged nursing home residents: a multi-center prevalence and correlational study. BMC Geriatr. 2017 Nov 13;17(1):263. doi: 10.1186/s12877-017-0655-5. PMID 29132305
- [Background] Kayser SA, Phipps L, VanGilder CA, Lachenbruch C. Examining Prevalence and Risk Factors of Incontinence-Associated Dermatitis Using the International Pressure Ulcer Prevalence Survey. J Wound Ostomy Continence Nurs. 2019 Jul/Aug;46(4):285-290. doi: 10.1097/WON.0000000000000548. PMID 31276451
- [Background] Minematsu T, Yamamoto Y, Nagase T, Naito A, Takehara K, Iizaka S, Komagata K, Huang L, Nakagami G, Akase T, Oe M, Yoshimura K, Ishizuka T, Sugama J, Sanada H. Aging enhances maceration-induced ultrastructural alteration of the epidermis and impairment of skin barrier function. J Dermatol Sci. 2011 Jun;62(3):160-8. doi: 10.1016/j.jdermsci.2011.03.005. Epub 2011 Mar 23. PMID 21498052
- [Background] Mugita Y, Koudounas S, Nakagami G, Weller C, Sanada H. Assessing absorbent products' effectiveness for the prevention and management of incontinence-associated dermatitis caused by urinary, faecal or double adult incontinence: A systematic review. J Tissue Viability. 2021 Nov;30(4):599-607. doi: 10.1016/j.jtv.2021.07.002. Epub 2021 Jul 13. PMID 34376333
- [Background] Musa MK, Saga S, Blekken LE, Harris R, Goodman C, Norton C. The Prevalence, Incidence, and Correlates of Fecal Incontinence Among Older People Residing in Care Homes: A Systematic Review. J Am Med Dir Assoc. 2019 Aug;20(8):956-962.e8. doi: 10.1016/j.jamda.2019.03.033. Epub 2019 May 23. PMID 31129021
- [Background] Nix DH. Validity and reliability of the Perineal Assessment Tool. Ostomy Wound Manage. 2002 Feb;48(2):43-6, 48-9. PMID 15382413
- [Background] Shin YS, Kim HJ, Moon NK, Ahn YH, Kim KO. The effects of uncoated paper on skin moisture and transepidermal water loss in bedridden patients. J Clin Nurs. 2012 Sep;21(17-18):2469-76. doi: 10.1111/j.1365-2702.2012.04160.x. PMID 22889444
- [Background] Sugama J, Sanada H, Shigeta Y, Nakagami G, Konya C. Efficacy of an improved absorbent pad on incontinence-associated dermatitis in older women: cluster randomized controlled trial. BMC Geriatr. 2012 May 29;12:22. doi: 10.1186/1471-2318-12-22. PMID 22642800
- [Background] Yeomans A, Davitt M, Peters CA, Pastuszek C, Cobb S. Efficacy of chlorhexidine gluconate use in the prevention of perirectal infections in patients with acute leukemia. Oncol Nurs Forum. 1991 Sep-Oct;18(7):1207-13. PMID 1945967
- See also: Incontinence-associated dermatitis: moving prevention forward — https://www.researchgate.net/publication/299365578_Incontinence-associated_dermatitis_moving_prevention_forward
- See also: The Impact of an Absorbent Underpad on the Prevention and/or Improvement of Incontinence Associated Dermatitis in Skilled Nursing Facility (SNF) Residents. — https://doi.org/10.1016/j.jamda.2015.12.089
- See also: IAD made easy. — https://woundsinternational.com/made-easy/iad-made-easy/